CLINICAL TRIAL: NCT01292278
Title: The Possible Role of Neuropeptide Y After Spontaneous Subarachnoid Hemorrhage
Brief Title: Constitution of Cerebrospinal Fluid and Blood Database/Specimen in Acute Stage of Subarachnoid Hemorrhage (aSAH) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Regensburg (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Karl-Michael Schebesch, Karl-Michael Schebesch, MD, University of Regensburg
Other Study IDs: CSF 06/179
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Subarachnoid Hemorrhage
Keywords: subarachnoid hemorrhage; cerebral vasospasm; neuropeptide Y; spontaneous; aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cerebrospinal fluid / serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- aSAH: consecutive patients with spontaneous or aneurysmal subarachnoid hemorrhage
- control group: no neurological disease but spinal anesthesia

SUMMARY:
Neuropeptide Y (NPY) may play a major role in the pathophysiology of aneurysmal subarachnoid hemorrhage (aSAH). To investigate the correlation of NPY in cerebrospinal fluid (CSF) and blood (serum) and the neurological outcome in the acute stage of aSAH.

DETAILED DESCRIPTION:
Evaluation of Neuropeptides in CSF and serum in SAH patients

ELIGIBILITY:
Inclusion Criteria:

* spontaneous or aneurysmal subarachnoid hemorrhage

Exclusion Criteria:

* age younger than 18 years or older than 70 years
* inflammatory disease
* history of former SAH
* no ventricular drainage

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: consecutive pts. with subarachnoid hemorrhage
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2006-01; Primary Completion 2015-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale | 2011-2016

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery Medical Center University of Regensburg, Regensburg, Germany